CLINICAL TRIAL: NCT02676687
Title: Supratotal Resection for Gliomas Within Noneloquent Areas: A Single Center Prospective Randomized Controlled Clinical Trial
Brief Title: Supratotal Resection for Gliomas Within Noneloquent Areas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Rong Hu, Associate Professor, Associate Chief Neurosurgeon, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Neurosurg02
Record Dates: First submitted 2016-01-29; First posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Glioma
Keywords: surgery, noneloquent area
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- total resection (Active Comparator): Removing the parenchyma until signal abnormalities on FLAIR-weighted MR / enhanced-weighted MR in adults with glioma
  Interventions: Procedure: total resection
- supratotal resection (Experimental): Extended removing the parenchyma at least 1cm beyond signal abnormalities on FLAIR-weighted MR / enhanced-weighted MR in adults with glioma
  Interventions: Procedure: supratotal resection

INTERVENTIONS:
Procedure: total resection — Removing the parenchyma until signal abnormalities on FLAIR-weighted MR / enhanced-weighted MR in adults with glioma
  Arms: total resection
Procedure: supratotal resection — Extended removing the parenchyma at least 1cm beyond signal abnormalities on FLAIR-weighted MR / enhanced-weighted MR in adults with glioma
  Arms: supratotal resection

SUMMARY:
Gliomas, especially high grade gliomas and diffuse low grade gliomas, are characterized by their infiltrative nature. Recently, a new conception of supratotal resection has been proposed. Given the lack of prospective supporting data, the correlation between supratotal resection and the survival of patients with glioma need to be established.

Therefore, the investigators aim to do a single center prospective randomized controlled clinical trial to assess the effect of supratotal resection at least 1 cm beyond the MR imaging-defined abnormalities on progression-free survival (PFS) of glioma.

DETAILED DESCRIPTION:
It has been demonstrated that an extensive resection (total or subtotal) significantly increases the overall survival in patients with gliomas. Yet, recent data have shown that conventional MR imaging underestimates the spatial extent of gliomas, since tumor cells were found to invade beyond MR imaging abnormalities. Thus, it is hypothesized that an extended resection with a margin beyond MR imaging-defined abnormalities-a "supratotal" resection-might improve the outcome of gliomas. However, the exact extent of supratotal resection remains unclear. Unnecessary removal of brain tissue that does not contain cancer cells can lead to neurological deficits that affect quality of life, such as impaired cognition, memory, and vision. Recently, studies from human specimens have shown that infiltrating glioma cells spread about 1cm beyond the gross and radiographic margins of the tumor. The investigators thereof propose to perform extended resection at least 1cm beyond the MRI defined margin might improve the outcome of patients with gliomas.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18-80 years with highly suspected (as assessed by study surgeon), newly diagnosed, untreated glioma
2. Tumor in noneloquent brain areas diagnosed by Head MRI, an eloquent areas is defined according to the recent UCSF (University of California, San Francisco) classification, including the sensor motor areas (precentral and postcentral gyri), perisylvian language areas in the dominant hemisphere (superior temporal, inferior frontal, and inferior parietal gyri), basal ganglia, internal capsule, thalamus, and visual cortex around the calcarine sulcus
3. Lesions located at least 1 cm far away from an eloquent area and important subcortical tracts such as pyramidal tract, uncinate fasciculus (preoperatively roughly estimated by MRI and DTI)
4. Individuals who can accept and complete Stupp regimen therapy after surgery
5. Karnofsky performance scale (KPS) 70 or more
6. All patients giving written informed consent.

Exclusion Criteria:

1. Individuals with age < 18 years or > 80 years
2. Tumors in eloquent areas, as well as tumors with long invasion (i.e., crossing the corpus callosum) and deep seated tumors (i.e., basal ganglia)
3. Recurrent gliomas after surgery (except needle biopsy)
4. Pregnancy or breast-feeding women
5. Unable to achieve imaging data
6. Inability to give written informed consent
7. KPS < 70
8. Heart insufficiency, lungs insufficiency, renal insufficiency, hepatic insufficiency, autoimmune diseases and other organ diseases with severe dysfunction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rates | 2 years

SECONDARY OUTCOMES:
Volume of resection | 3 days
Karnofsky performance scale (KPS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rong Hu, Ph.D, Principal Investigator — Southwest Hospital, China; Hua Feng, Ph.D, Principal Investigator — Southwest Hospital, China
Locations (1):
- Department of Neurosurgery , Southwest Hospital, Third Military Medical University,, Chongqing, China

IPD SHARING:
Plan to Share IPD: No